CLINICAL TRIAL: NCT05479344
Title: Personal and Environmental Correlates of Problematic Internet and Smartphone Use
Brief Title: My Journey: A Brief Contextual Behavioural Intervention Based on Meaning and Connection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, LI Yumei, Principal Investigator, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-22-CIR5-1
Record Dates: First submitted 2022-07-22; First posted 2022-07-29 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Social Media Addiction; Internet Gaming Disorder; Smartphone Addiction; Quality of Life; Psychological Distress
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contextual Behavioural Intervention Based on Meaning and Connection (Experimental): The current intervention involves the identification of strengths (the first week, 90 minutes of intervention), the perception of the meaning in life (the second week, 90 minutes of intervention), the learning of strategies to develop plan (the third week, 90 minutes of intervention), and the understanding of emotion regulation strategies (the fourth week, 90 minutes of intervention).
  Interventions: Behavioral: A Brief Contextual Behavioural Intervention Based on Strengths, Meaning, Hope and Connection
- Waiting list group (Other): The waiting list group will receive the same intervention at the end of the 3-month follow-up test.
  Interventions: Behavioral: A Brief Contextual Behavioural Intervention Based on Strengths, Meaning, Hope and Connection

INTERVENTIONS:
Behavioral: A Brief Contextual Behavioural Intervention Based on Strengths, Meaning, Hope and Connection — The intervention strategy combines acceptance and commitment therapy, contextual behavioral science, and positive psychology interventions (strengths, meaning, hope) in the form of a single intervention set (each topic is a single 90-minute intervention, four single intervention combinations).

SUMMARY:
The present study will explore the underlying mechanisms of problematic Internet and smartphone use by focusing on how and when environmental factors affect the positive psychological intervention factors. Hence, the present study will provide scientific empirical evidence to design and formulate follow-up intervention strategies.

Aims:

I. Apply the dynamic system model of addictive behavior execution in Chinese adolescents with problematic Internet and smartphone use and use longitudinal data to track and explore the underlying mechanisms of environmental factors and personal factors on problematic Internet and smartphone use.

II. Identify positive psychological intervention factors that effectively prevent and reduce problematic Internet and smartphone use according to the interview and provide empirical evidence for other intervention designs.

III. Conducting a positive psychological intervention in an adolescent population to verify the protective effect of positive psychology factors on problematic Internet and smartphone use.

Hypotheses:

I. Environmental factors (e.g., child abuse and trauma, parenting behaviors, teachers' encouragement, peer support) will affect the problematic Internet and smartphone use through personal characteristics (e.g., meaning in life); II. The effect of environmental factors on problematic Internet and smartphone use through personal characteristics will be moderated by other positive psychological intervention factors (e.g., character strengths); III. Positive psychological intervention (e.g., meaning-based intervention, strengths-based intervention) is an effective intervention strategy to prevent and reduce problematic Internet and smartphone use.

DETAILED DESCRIPTION:
Problematic Internet and smartphone use are a psychosocial phenomenon in which individuals pay too much attention to and rely on the Internet, negatively affecting their mental and physical health, lives, and work. Many studies have shown that problematic Internet and smartphone use can bring adverse psychological effects (e.g., depression, anxiety, and negative emotions) and unfavorable physiological conditions (e.g., poor sleep quality and memory loss). The negative psychological and physiological effects can result in adverse academic and work performance outcomes. Many existing studies mainly explore the underlying mechanism of problematic Internet and smartphone use from personal factors such as mental health, metacognition, coping strategies, personality traits, motivation, and attachment styles. However, more and more studies have begun to focus on the effects of environmental factors, such as peer relationships and parenting styles, on problematic Internet and smartphone use. To fill the literature gaps, formulate effective preventive and remedial interventions, and explore whether, when, and how environmental factors (e.g., child abuse and trauma, parenting behaviors, teachers' encouragement, and peer support) affect problematic Internet and smartphone use is crucial.

The previous psychological interventions for problematic Internet and smartphone use focused on cognitive behavioral therapy, sand-play therapy, family programming, group programming, counseling programming, and educational programming. Different types of interventions reduced the severity of problematic Internet and smartphone use to varying degrees. However, the existing intervention strategies ignore the perspective of positive psychology. In the country, some scholars proposed to discuss the self-regulation of addicts from the perspective of positive psychology and especially proposed a meaning-centered approach as an essential supplement to mainstream addiction therapy. Besides, some scholars have also noticed the role of positive psychological intervention factors, such as meaning in life and the formation and development of problematic Internet and smartphone use. Therefore, exploring the positive psychological intervention factors, especially the meaning in life and the construction and development of problematic Internet and smartphone use, is the starting point for developing evidence-based intervention strategies.

According to the Dynamic System Model of Developmental Psychopathology and the Interaction of Person-Affect-Cognition-Execution model, the present study will explore the underlying mechanisms from environmental factors (e.g., child abuse and trauma, parenting behaviors, teachers' encouragement, peer support) to problematic Internet and smartphone use by testing the mediator role and moderator role of personal factors (e.g., the meaning of life, social media flow), predominantly positive psychological intervention factors (e.g., character strengths). Therefore, the present study integrated positive psychological intervention factors into the dynamic system model of addictive behavior execution and applies it to explore the formation and development mechanisms of problematic Internet and smartphone use (see Figure 1 and Figure 2). In addition, this study will implement an interview and meaning-centered intervention program among middle school students to validate the validity of the dynamic system model of addictive behavior execution from the interpretation of qualitative material and intervention practices.

Given the research variables' diversity and complexity, the present study intends to include at least 500 adolescents over 12 years of age. The present study uses convenience and snowball sampling in mainland China and Hong Kong. The present study will also invite participants to accept longitudinal tracking. Participants willing to participate in the subsequent two surveys will provide their contact information. Before the research, the parents' and children's online informed consent forms will be obtained for the minors' sample. This questionnaire survey was completed in the preliminary stage of this study (approved: 2020-21-CIR8-3), and the intervention directions and techniques for problematic Internet and smartphone use were determined based on the questionnaire survey results.

Semi-structured Interviews:

The investigators will use a method of semi-structured interviews with open-ended questions to collect data. Individual interviews, lasting between 45 and 60 minutes, will be conducted and recorded. All participants should provide consent to participate before being interviewed. The interviews were conducted in Mandarin. All the materials used in the study (e.g., the recruitment information and questionnaires) were presented in Chinese. Thirty adolescents will be recruited to participate in the interviews.

Randomized Controlled Trial:

The investigators will pilot test the proposed meaning-focused intervention using a randomized (1:1) parallel-group controlled, single-blind trial in middle school students. The middle school collaborators will help launch the advertisement regarding this study, brief potential participants, prescreen potential participants according to recruitment criteria, and recruit participants using the opportunity sampling method. The participants' written informed consent will be obtained before conducting the intervention. One hundred adolescents will be recruited to participate in a randomized controlled trial. Four sessions will be delivered to the intervention group 1 week apart, with around 90 minutes per session.

Descriptive analysis and latent profile analysis will be adopted to present the overall situation of the research sample; psychology measurement attributes of the measures will be tested using confirmatory factor analysis; the correlation and regression analysis will be used to explore the relationships between environmental factors, personal factors, and problematic Internet and smartphone use. The structural equation modeling will be conducted to verify the mediator or moderator roles of positive psychological intervention factors in the relationship between environmental factors and problematic Internet and smartphone use.

ELIGIBILITY:
Inclusion Criteria:

1. Children or adolescents with experience in using technology.
2. Older than 12 years and younger than 20 years.
3. Native Chinese speakers.

Exclusion Criteria:

1. Young people with no experience in using technology.
2. Aged under 12 or over 20.
3. Non-native speakers of Chinese.
4. People who have undergone similar interventions within the past year.
5. Persons with major mental or physical illnesses.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change of Problematic Social Media Use | baseline, week 5, 3-month follow up
  The 6-item Bergen Social media Addiction Scale will measure the severity of problematic social media use. Bergen Social media Addiction Scale is a self-report measure designed to assess the symptoms of problematic social media use, with a higher total score suggesting more severe problematic use symptoms. Scores range from 6 to 30.
Change of Problematic Smartphone Use | baseline, week 5, 3-month follow up
  The 6-item Smartphone Application-Based Addiction Scale will measure the severity of problematic smartphone use. Smartphone Application-Based Addiction Scale is a self-report measure designed to assess the symptoms of problematic smartphone use, with a higher total score suggesting more severe problematic use symptoms. Scores range from 6 to 36.
Change of Internet Gaming Disorder | baseline, week 5, 3-month follow up
  The 9-item Internet Gaming Disorder Scale-Short Form will measure the severity of internet gaming. Internet Gaming Disorder Scale-Short Form is a self-report measure designed to assess the symptoms of internet gaming disorder, with a higher total score suggesting more severe internet gaming symptoms. Scores range from 9 to 45.
Change of Depression and Anxiety Symptoms | baseline, week 5, 3-month follow up
  Anxiety and depressive symptoms will be measured by the 4-item Patient Health Questionnaire for Depression and Anxiety (PHQ-4). PHQ-4 is a self-report measure designed to assess the severity of depression and anxiety symptoms, with a higher total score suggesting higher levels of depression and anxiety symptoms. Scores range from 0 to 12.

SECONDARY OUTCOMES:
Change of Meaning in Life | baseline, week 5, 3-month follow up
  The 24-item State of Meaning in Life Scale will be used to measure the meaning in life. State of Meaning in Life Scale is a self-report measure designed to assess the six dimensions (need for meaning, meaning avoidance, meaning anxiety, meaning confusion, search for meaning, and presence of meaning) of meaning in life, with a higher mean score suggesting a higher levels of that state of meaning in life. Scores range from 1 to 7.
Change of Difficulties in Emotion Regulation | baseline, week 5, 3-month follow up
  The 18-item Difficulties in Emotion Regulation Scale Short Form (DERS-SF) will be used to measure the difficulties in regulating emotions. DERS-SF is a self-report measure designed to six factors of difficulties in regulating emotions (regulation strategies, non-acceptance of emotional responses, impulse control difficulties, goal-directed difficulties, awareness difficulties, emotional clarity difficulties), with a higher total score denoted a higher level of difficulties in regulating emotions. Scores range from 18 to 90.

CONTACTS AND LOCATIONS:
Overall Officials: Yumei LI, Principal Investigator — Department of Social & Behavioural Sciences, City University of Hong Kong
Locations (1):
- Chongqing Datong High School, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study dataset will contain identifiable information about minors, and therefore ethical clearance requires that no one other than our study team have access to the data collected in this study.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT05479344/ICF_000.pdf